CLINICAL TRIAL: NCT03845829
Title: Left Subclavian Artery Reconstruction With Laser-assisted Fenestration During the Procedure of Thoracic EndoVascular Aortic Repair for Type B Aortic Dissection
Brief Title: LSA Reconstruction With Laser Fenestration During the TEVAR
Acronym: LLTEVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Kaichuang Ye, MD, PhD, Department of Vascular Surgery, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAL01
Record Dates: First submitted 2019-01-29; First posted 2019-02-19 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Type B Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with TBAD treated with TEVAR (Experimental): In situ laser assisted fenestration for the left subclavian artery during the TEVAR procedure for TBAD.
  Interventions: Procedure: In situ laser assisted fenestration

INTERVENTIONS:
Procedure: In situ laser assisted fenestration — In situ laser assisted fenestration for the left subclavian artery during the procedure of TEVAR for type B aortic dissection

SUMMARY:
This study aims to evaluate the feasibility, effectiveness, and safety of in-situ laser-assisted fenestration on the left subclavian artery during the procedure of thoracic artery endovascular repair

DETAILED DESCRIPTION:
This study is a single-arm, prospective study. All patients with type B aortic dissection (TBAD) present with the proximal tear site located approximately close to the left subclavian artery and a reconstruction of the left subclavian artery is necessary are included in the present study. During the procedure of thoracic artery endovascular repair (TEVAR), the left subclavian artery will be reconstructed with laser-assisted fenestration and the fenestrated stent will be covered stents (fluency, viabhan, lifestream).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female over 18 years of age;
* Type B Aortic Dissection;
* The left subclavian artery should be reconstructed during the TEVAR procedure.
* Patient is willing to provide informed consent and comply with the required follow up visits, testing schedule and medication regimen;

Exclusion Criteria:

* Life expectancy of < 5 years;
* Patients need open surgery repair for the aortic diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaichuang Ye, MD, PhD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Kaichuang Ye, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng Z, Liang S, Zhang R, Qiu P, Yin M, Liu G, Liu X, Lu X, Ye K. Left Subclavian Artery Revascularization With In Situ Laser Fenestration During Thoracic Endovascular Aortic Repair for Acute Complicated or High-Risk Type B Aortic Dissection: Results of the LLTEVAR Trial. J Am Heart Assoc. 2025 Dec 16;14(24):e041720. doi: 10.1161/JAHA.125.041720. Epub 2025 Dec 10. PMID 41368828

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patient was excluded in this study when enrolled.
Groups:
- Patients With Complicated and High-risk TBAD Treated With TEVAR: In situ laser assisted fenestration for the left subclavian artery during the TEVAR procedure for TBAD.
  In situ laser assisted fenestration: In situ laser assisted fenestration for the left subclavian artery during the procedure of TEVAR for type B aortic dissection
Period: Overall Study
Arm/Group | Patients With Complicated and High-risk TBAD Treated With TEVAR
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With TBAD Treated With TEVAR
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 100
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China: Shanghai ninth people's hospital, Shanghai Jiaotong University School of Medicine | 48
  China: Shanghai third people's hospital, Shanghai Jiaotong University School of Medicine | 27
  China: Taizhou Municipal hospital, Taizhou, Zhejiang | 13
  China: Zhoupu Hospital, Pudong, Shanghai | 6
  China: Fengcheng Hospital, Fengxian, Shanghai | 6
smoking [Count of Participants; unit: Participants] | 38
BMI >25 [Count of Participants; unit: Participants] | 29
Comorbidity [Number; unit: participants]
  Hypertension | 90
  Diabetes | 8
  Ischemia heart disease | 8
  Cerebrovascular disease | 7
  Congestive heart failure | 1
  Chronic obstructive pulmonary disease | 11
  Chronic kidney disease | 6
  Chronic renal artery occlusion | 2
  Acute mesenteric ischemia | 3
  Acute limb ischemia | 6
Time from onset of symptoms to procedure [Count of Participants; unit: Participants]
  Hyperacute stage (<24h) | 26
  Acute stage (24h-14d) | 52
  Subacute stage (>14d) | 22
Aortic dissection acuity [Count of Participants; unit: Participants]
  Complicated | 18
  High risk | 82

OUTCOME MEASURES:

1. Primary Outcome: Freedom From All-cause Reintervention, All-cause Mortality and Major Adverse Events Within 30 Days After Procedure
Description: The primary safety endpoint was freedom from major adverse events within 30 days after procedure. The major adverse events included mortality, stroke, myocardial infarction, rupture, paraplegia, type Ia endoleak, major bleeding, acute kidney injury, limb ischemia, bowel ischemia, retrograde dissection, stent-induced new entry (SINE), access site complications and unplanned reinterventions.
Time Frame: within 30 days after procedure
Population: The primary safety endpoint was 84% (84/100), with 19 events occurring in 16 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Complicated and High-risk TBAD Treated With TEVAR
Number analyzed (Participants) | 100
Participants | 84

2. Secondary Outcome: Aortic Disease Related Mortality
Description: the incident of death associated with aortic disease.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Complicated and High-risk TBAD Treated With TEVAR
Number analyzed (Participants) | 100
Participants | 0

3. Secondary Outcome: Incidence of Endoleak Within 12 Months After Procedure
Description: During the follow up of 12 months after procedure, the total incidence of endoleaks.
  Type Ia endoleak is a perigraft leak at the proximal edge of the stent graft that allows continued antegrade flow into the false lumen through the primary entry tear. Type Ib endoleak is a distal perigraft leak caused by a tear in the intimal membrane adjacent to the distal edge of the endograft (distal stent graft-induced new entry, SINE). Type II endoleak is continued retrograde false lumen perfusion through an arch branch (eg, left subclavian artery as demonstrated in the illustration) or intercostal or bronchial artery. Type R endoleak is antegrade flow from the true lumen to the false lumen through septal, visceral, or distal fenestrations.
Time Frame: 12 months
Population: all types of endoleak during the follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Complicated and High-risk TBAD Treated With TEVAR
Number analyzed (Participants) | 100
Participants
  R endoleak | 2
  II endoleak | 2
  Ib endoleak | 4
  Ia endoleak | 1

4. Secondary Outcome: Technical Success Rate During the Procedure
Description: Technical success of successful TEVAR procedure and the in-situ laser-assisted fenestration for LSA revascularization.
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Complicated and High-risk TBAD Treated With TEVAR
Number analyzed (Participants) | 100
Participants | 98

5. Secondary Outcome: Patency Rate of Branches Stents 12 Months After Procedure
Description: Patency rate (less than 50% in-stent-restenosis) of the subclavian artery stents 12 months after procedure.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Complicated and High-risk TBAD Treated With TEVAR
Number analyzed (Participants) | 100
Participants | 98

ADVERSE EVENTS:
Time Frame: with 30 days after procedure.
Description: The major adverse events included mortality, stroke, MI, rupture, paraplegia, type Ia endoleak, major bleeding, AKI, limb ischemia, bowel ischemia, retrograde dissection, SINE, access site complications and unplanned reinterventions, which was referred to intervention for major adverse events, included surgical repair for ascending aortic pathologies, coronary artery stenting, embolism for type Ia endoleak, additional proximal or distal aortic stents deployment, intervention for access sites.
Arm/Group | Patients With Complicated and High-risk TBAD Treated With TEVAR
All-Cause Mortality (participants affected / at risk) | 2/100
Serious Adverse Events (participants affected / at risk) | 16/100
Other Adverse Events (participants affected / at risk) | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Complicated and High-risk TBAD Treated With TEVAR (N=100)
Stroke (Cardiac disorders) | 4 (4)
Myocardial infarction (Cardiac disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Mesenteric ischemia (Gastrointestinal disorders) | 1 (1)
Ia endoleak (Vascular disorders) | 5 (5)
Spinal cord ischemia (Nervous system disorders) | 1 (1)
Retrograde dissection (Vascular disorders) | 1 (1)
Retrograde IMH (Vascular disorders) | 1 (1)
Access site pseudoaneurysm (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03845829/Prot_SAP_000.pdf